CLINICAL TRIAL: NCT03848663
Title: Remapping the Visual Field to Aid Reading With Central Scotomas
Brief Title: Visual Remapping to Aid Reading With Field Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMAP002
Record Dates: First submitted 2019-01-28; First posted 2019-02-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Age-related Macular Degeneration
Keywords: Scotoma; Remapping; Reading; Low vision; Visual aid
MeSH Terms: conditions — Macular Degeneration; Scotoma; Vision, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with scotoma (Experimental): No remapping (control condition), traditional remapping, personalized remapping
  Interventions: Behavioral: Traditional Remapping; Behavioral: Personalized Remapping
- Normally sighted with artificial scotoma (Active Comparator): No remapping (control condition), traditional remapping, personalized remapping
  Interventions: Behavioral: Traditional Remapping; Behavioral: Personalized Remapping

INTERVENTIONS:
Behavioral: Traditional Remapping — Shifting text outside of scotoma
Behavioral: Personalized Remapping — Shifting text based on individual letter-based perimetry

SUMMARY:
Reading performance in patients with Central Vision Loss and age matched controls with artificial scotomas will be measured with and without different kinds of remapping of missing text to different parts of the visual field.

DETAILED DESCRIPTION:
Following initial characterization of their visual field loss, the participant's performance in reading tasks will be measured with and without remapping. Tasks will include reading groups of random letters, words, simple sentences, and "natural" text from the environment (taken from phone apps, signage, etc). Different kinds of remappings will be used by participants, including traditional and personalized remapping. For control observers, differently shaped artificial scotomas will be used.

Participants interested in the study will be brought in for an initial visit. All participants will be administered the MMSE. Observers who pass the criteria for the study will then have the remainder of the procedures described to them verbally prior to undergoing the remainder of the consent process (see below). Participants will then undergo a standard exam at the UMN eye clinic, if they have not had one within the last month.

Participants will then have their scotomas mapped using a microperimeter housed in the psychology department to give size and shape information. Additional perimetry may also be conducted using either of the two displays (either HMD or desk mounted computer monitor) we have developed. Here, patients will be asked to fixate at a spot on screen and identify visual stimuli presented at different regions of the screen. The size and locations of visual stimuli patients were unable to identify will provide the size and location of the scotoma. Another additional manual perimetry protocol may be conducted as well. This would involve asking subjects to fixate at the center of a tangent screen, and asking them to identify dots temporarily presented on the screen by the researcher using a laser pointer. The locations of dots that patients are unable to identify will provide the size and location of the scotoma. The location and extent of each eye's scotoma and PRL will be used as software inputs on either device. Perimetry using one or all of the methods above will be performed until acceptable information about the scotoma extent and location is obtained.

In a second visit, participants will perform the visual tasks that are used as the basis of their personalized remapping, letter perimetry. Participants will first view and report three randomly selected horizontally arranged letters placed at different locations in the visual field. This letter perimetry task will take about 40 min and will cover a large part of the visual field.

Participants will then read single words whose letters have been displaced from horizontal in various ways that comprise candidate remappings generated on the basis of the letter perimetry results. This personalization test will take about 40 minutes, and will find a good remapping strategy for the individual. Subjects will then be introduced to the reading tasks that comprise the remainder of the study

In 6 additional sessions, participants will perform various reading tasks using different remappings. In all of these, text will be displayed on the screen, and the task is simply to read aloud what was presented. Two sessions will involve reading single words, one session will involve reading strings of 3 letters that are not arranged horizontally, two sessions will involve reading short sentences, and one session will involve reading naturalistic text (from phone apps, signage, menus, etc). In all sessions, some reading will be with remapping, some will be without. Both traditional and personalized remapping will be used.

In all these sessions, the eye tracker will be calibrated to participants' individual head and eye position. This will involve fixating at different points on the device screen (HMD or desk-mounted) as the eye is imaged by the eye trackers. This may take up to 45 minutes in the initial session, if various combinations of head and eye positions are required for the eye trackers to work well. But once completed, calibration is much faster in subsequent sessions. Quick perimetry validation may also be conducted in each session.

Throughout all testing, patients will be asked if they feel any discomfort, and will be able to take a break or quit testing at any point.

Including the initial visit, testing for any given patient is anticipated to last no more than eight sessions over eight weeks. Enrolling participants, testing, and data analysis for all participants is anticipated to take five years from the date of enrollment of the first participant.

ELIGIBILITY:
Inclusion Criteria:

1. 16 years or older
2. Central vision loss of at least 5 deg diameter, including the fovea, from bilateral central scotomas
3. Stable fixation (+/- 1 deg) using their PRL.
4. No cognitive impairment as indicated by a Mini-Mental State Examination (MMSE).
5. Satisfactory calibration achievable using eye tracker

Exclusion Criteria:

1. Central vision loss of less than 5 deg diameter; scotomas that do not cover the fovea; unilateral scotomas
2. Poor fixation (worse than+/- 1 deg) using their PRL.
3. Cognitive impairment as indicated by a Mini-Mental State Examination (MMSE).
4. Satisfactory calibration not achievable using eye tracker

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Reading Speed for Individual Words | Measured during third visit- each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  How quickly participants can correctly read displayed text
Reading Speed for Sentences | Measured during fourth visit- each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  How quickly participants can correctly read displayed text
Reading Speed for Natural Text Samples | Measured during fifth visit; each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  How quickly participants can correctly read displayed text
Reading error rate for Individual Words | Measured during third visit; each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  How many mistakes participants make
Reading error rate for Sentences | Measured during fourth visit; each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  How many mistakes participants make
Reading error rate for Natural Text Samples | Measured during fifth visit; each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  How many mistakes participants make

SECONDARY OUTCOMES:
Eye fixation quality for words | Measured during third visit; each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  Variance of x and y eye position coordinates computed during fixation periods while reading
Eye fixation quality for sentences | Measured during fourth visit; each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  Variance of x and y eye position coordinates computed during fixation periods while reading
Eye movement quality for sentences | Measured during fourth visit
  Number off leftward (regressive) eye movements during sentence reading
Eye fixation quality for natural text samples | Measured during fifth visit; each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  Variance of x and y eye position coordinates computed during fixation periods while reading
Eye movement quality for natural text samples | Measured during fifth visit; each visit is one day only and this measure refers to data gathered during a < 1 hr long reading session during that day
  Number off leftward (regressive) eye movements during natural text reading

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Engel, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Perimetry, psychophysical and eye-tracking data will be deidentified upon acquisition, and indexed using only a subject code. These data will be stored on a secure server for sharing upon request by a PI of a research team. We will offer psychophysical and eye tracking data along with appropriate metadata specifying details of the test (remapping used, stimulus protocol, etc) and data format.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Once results are published.
Access Criteria: Research group.